CLINICAL TRIAL: NCT03813095
Title: Nanoencapsulated Cannabidiol Time Released Capsules Targeted to Reduce Cravings in the Treatment of Opioid Addiction
Brief Title: Exploratory Dose Ranging Study Assessing APH-1501 for the Treatment of Opioid Addiction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aphios (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APH-1501
Record Dates: First submitted 2019-01-14; First posted 2019-01-23 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Addiction; Opioid Dependence; Opioid Withdrawal
Keywords: Addiction; Cannabis; Substance Use; Opioids: Harmful Use; Cocaine; Neurotransmitter Uptake Inhibitors; Analgesics; Mental Disorders; Narcotics; Cannabidiol
MeSH Terms: conditions — Behavior, Addictive; Opioid-Related Disorders; Marijuana Abuse; Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- APH-1501 400mg (Experimental): Nano-encapsulated for oral delivery. The study is planned for patients to receive APH 1501 400mg BID( twice daily) for 28 days.
  Interventions: Drug: APH-1501
- APH-1501 600mg (Experimental): Nano-encapsulated for oral delivery. The study is planned for patients to receive APH 1501 600mg BID ( twice daily) for 28 days.
  Interventions: Drug: APH-1501
- APH-1501 800mg (Experimental): Nano-encapsulated for oral delivery. The study is planned for patients to receive APH 1501 800mg BID ( twice daily) for 28 days.
  Interventions: Drug: APH-1501
- Placebo Comparator: Placebo (Placebo Comparator): Nano-encapsulated for oral delivery. The study is planned for patients to receive a placebo dose BID ( twice daily) for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APH-1501 — The investigational drug product APH-1501 is CBD encapsulated in biodegradable polymer nanospheres, is a lyophilized powder intended for oral administration.
  Arms: APH-1501 400mg; APH-1501 600mg; APH-1501 800mg
Drug: Placebo — The placebo is a sterile pyrogen free lyophilized powder identical in appearance to the experimental drug product.
  Arms: Placebo Comparator: Placebo

SUMMARY:
The purpose of this study is determine the safety, efficacy and tolerability of a novel drug APH-1501 as a pharmacotherapy for Opioid Dependence. The investigators will evaluate the safety of escalating doses APH-1501.

DETAILED DESCRIPTION:
This is a Phase 2a Exploratory Pilot study assessing the efficacy, immunogenicity and pharmacology of APH-1501, Cannabidiol (CBD), a unique, bioactive component of marijuana, in reducing early attrition and improving outcome in opioid-dependent individual in adults diagnosed with an opioid addiction, ages 21-55 years of age. Subjects will be randomized into 4 groups receiving APH-1501 or placebo over a 30 day period that includes a regimen of reformulated 400, 600 or 800 mg/m2 APH 1501 or placebo. This trial will target opioid-dependent patients who have completed detoxification and are in a treatment facility. During the trial period, participants will be given APH-1501 twice a day for 30 days. Given prior evidence based research on CBD there should be minimum to no side effects to taking APH 1501. The overarching research question for the study is the efficacy of APH 1501, pharmaceutical-grade CBD (>98.5% and < 0.3% Δ9-THC) for clinical use in the treatment of opioid addiction.

This is an intervention model design with three treatment groups, parallel assignment. This study is designed for sufficient time in between dose escalations to allow for interim analysis of safety and tolerability data to be considered for the safest approach to assess the effects of the compound as a therapeutic agent. Randomization will be stratified by the Diagnostic and Statistical Manual (DSM)_V diagnosis taking into account any co-morbid features or dual diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 21 to 55 Years (Adult)
* Sexes Eligible for Study: All
* Accepts Healthy Volunteers: No
* Meets DSM-V criteria with a Substance Use Disorder
* Meets protocol-specified criteria for qualification and contraception
* Must consent to random assignment, and be willing to commit to medication ingestion.
* Is willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff;
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding);
  3. the analysis of results
* Individuals with clinically significant medical disorders or lab abnormalities.
* History of cardiovascular events, head trauma or seizures
* Use of any psychoactive drug or medication at any time of study enrollment and participation
* Having taken any opioid medication in the last 14 days
* Concomitant use of psychotropic medications, with the exception of stable doses (defined as no dosing adjustments in the past two months) of non-monoamine oxidase inhibitor (MAO-I) (antidepressants, non-benzodiazepine anxiolytics, and Attention Deficit -Hyperactivity Disorder(ADHD) medications.
* Pregnant or breastfeeding
* Not using appropriate contraceptive measures ( hormonal, Nuvo-ring, Depo-Provera, IUD) or other barrier protection.
* Psychiatric condition as defined by the DSM-V - Lifetime history of DSM-5 Bipolar I or II Disorder, Schizophrenia or other psychotic disorder. Stably treated Major Depressive Disorder (MDD), Dysthymia, Generalized Anxiety Disorder (GAD), Social Phobia, and Specific Phobia diagnoses are acceptable (i.e. same dose of medication has been prescribed for at least 2 months prior to screening and no changes in current medication expected during course of the trial).
* Hypersensitivity to cannabinoids
* Suicidal ideation or behavior within the past 6 months. Subjects who are believed to be at suicidal or homicidal risk (answers 'yes' on questions 4 or 5 of C-SSRS) will be referred for assessment by a qualified mental health professional.
* Individuals taking an investigational agent within the last 30 days before baseline visit.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
[Safety] Incidence of Treatment Emergent Adverse Effects | Baseline through 30 days post final treatment dose up to day 60
  Number of patients experiencing treatment emergent Adverse Effects(AE's) and Serious Adverse effects(SAE's) during treatment and follow-up. Patients will be asked to complete the Systematic Assessment for Treatment Emergent Events (SAFTEE)
  The SAFTEE is a questionnaire that rates the current severity of a wide range of somatic, behavioral and affective symptoms in general and specific inquiry formats. It is designed to report adverse health events. Contains ~ 25 detailed questions that systematically address 29 body systems. Responses are rated on five levels of severity.
[Tolerability] Pharmacokinetics of APH-1501 | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes 240 minutes, 480 minutes post administered dose
  Blood draws to determine the cannabidiol peak plasma concentration (Cmax).
[Tolerability] Pharmacokinetics of APH-1501 | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes 240 minutes, 480 minutes post first administered dose.
  Blood draws to determine the cannabidiol time to reach peak serum concentration (Tmax).
[Tolerability] Pharmacokinetics of APH-1501 | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes 240 minutes, 480 minutes post first administered dose.
  Blood draws to determine the cannabidiol time to derermine serum half life (1/2).

SECONDARY OUTCOMES:
Vital signs | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes 240 minutes, 480 minutes, post first administered dose.
  Change in Blood pressure - diastolic & systolic (in mmHg).
Vital signs | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes 240 minutes, 480 minutes, post first administered dose.
  Change in Heart Rate( beats per minute).
Vital signs | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes 240 minutes, 480 minutes, post first administered dose.
  Change in Respiratory (in breaths per minute).
Vital signs | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes 240 minutes, 480 minutes, post first administered dose.
  Change in Temp ( in degrees Farenheit).
Vital signs | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes 240 minutes, 480 minutes, post first administered dose.
  Change in O2 saturation.
Vital signs | Baseline, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 120 minutes, 180 minutes 240 minutes, 480 minutes, post first administered dose.
  Change in Electrocardiogram (ECG). ( P Wave and QRS Complex)
Vital signs | Day 7,14,21,28 and 60 for followup.
  Change in Blood pressure(in mmHg) diastolic and Systolic.
Vital signs | Day 7,14,21,28 and 60 for followup.
  Change in Heart Rate( beats per minute).
Vital signs | Day 7,14,21,28 and 60 for followup.
  Change in Respiratory (in breaths per minute).
Vital signs | Day 7,14,21,28 and 60 for followup.
  Change in Temp ( in degrees Farenheit).
Vital signs | Day 7,14,21,28 and 60 for followup.
  Change in O2 saturation.
Vital signs | Day 7,14,21,28 and 60 for followup.
  Change in Electrocardiogram ( EKG) P Wave and QRS Complex
Anxiety | Baseline, weeks 1-4 and 1 week post final dose.
  Anxiety Assessment using the Beck Anxiety Inventory ( BAI) . The BAI is a self-report measure of anxiety. The total score is calculated by finding the sum of the 21 items. Score of 0-21 = low anxiety Score of 22-35 = moderate anxiety Score of 36 and above = potentially concerning levels of anxiety
Changes in levels of physiological stress | Baseline through 30 days post final treatment dose up to day 60
  Measure salivary cortisol levels
Visual Analog Scale for Craving | Baseline, weeks 1-4 and 30 days post final treatment up to day 60
  Changes and potential variations in cue-induced craving will be monitored and measured.
Clinical Opiate Withdrawal Scale ( COWS) | Baseline, weeks 1-4 adn 30 days post final treatment up to day 60
  Changes and variations in common signs and symptoms of opiate withdrawal will be measured and monitor over time.

IPD SHARING:
Plan to Share IPD: No